CLINICAL TRIAL: NCT03459157
Title: Access to Pre-exposure Prophylaxis for Men Who Have Sex With Men: Acceptability and Feasibility in Community-based Clinics in West Africa (CohMSM-PrEP)
Brief Title: Access to PrEP for MSM: Acceptability and Feasibility in Community-based Clinics in West Africa (CohMSM-PrEP)
Acronym: CohMSM-PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Expertise France (Other); Université Montpellier (Other); SESSTIM (IRD, Inserm, Université Aix-Marseille) (Unknown); Coalition Internationale Sida (Other); Institut de Médecine Tropicale, Anvers, Belgique (Unknown); ARCAD-SIDA MALI (Other); Association African Solidarité (Other); Centre de Recherche Internationale pour la Santé, Université de Ouagadougou (Unknown); Espace Confiance, Côte d'Ivoire (Other); Espoir Vie-Togo - ONG (Other); Laboratoire BIOLIM, Université de Lomé (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12369 CohMSM-PrEP
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: HIV/AIDS
Keywords: HIV infection; Men who have sex with men; Pre-exposure prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Homosexuality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV prevention package including PrEP (Other)
  Interventions: Drug: HIV prevention package including PrEP

INTERVENTIONS:
Drug: HIV prevention package including PrEP — All MSM enrolled will benefit from a comprehensive HIV prevention package including quarterly clinical examinations, screening and treatment of STIs, screening of HIV, PrEP (TDF 300 mg + FTC 200 mg), daily or on-demand, according the participant's choice, immunisation against hepatitis B, individualised peer-led support (for adherence and prevention), group discussions, condoms, and lubricants.

SUMMARY:
This demonstration project will assess the acceptability and feasibility of pre-exposure prophylaxis (PrEP) for men who have sex with men (MSM) as part of a comprehensive HIV prevention package in community-based clinics in West Africa.

An interventional, open label, multidisciplinary and multicentre cohort study will be performed in Burkina Faso, Côte d'Ivoire, Mali, and Togo.

All MSM enrolled will benefit from a comprehensive HIV prevention package including quarterly clinical examinations, screening and treatment of STIs, screening of HIV, PrEP (daily or on-demand, according the participant's choice), immunisation against hepatitis B, individualised peer-led support (for adherence and prevention), group discussions, condoms, and lubricants.

DETAILED DESCRIPTION:
This demonstration project will assess the acceptability and feasibility of pre-exposure prophylaxis (PrEP) for men who have sex with men (MSM) as part of a comprehensive HIV prevention package in community-based clinics in West Africa.

The specific objectives are to assess the acceptability of PrEP, the adherence to PrEP and to quarterly HIV testing, the safety of daily and on-demand use of TDF/FTC, the impact of PrEP on the other prevention strategies, the incidence of sexually transmitted infections (STIs) on PrEP, the "real life" effectiveness of PrEP use and treatment-related resistance, and the cost and cost-effectiveness of PrEP.

This interventional, open label, multidisciplinary and multicentre cohort study will be performed in Burkina Faso, Côte d'Ivoire, Mali, and Togo.

All MSM enrolled will benefit from a comprehensive HIV prevention package including quarterly clinical examinations, screening and treatment of STIs, screening of HIV, PrEP (daily or on-demand, according the participant's choice), immunisation against hepatitis B, individualised peer-led support (for adherence and prevention), group discussions, condoms, and lubricants.

These activities will be performed by community-based organisations which are pioneer in the fight against HIV, especially in MSM. The study will have a total duration of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Male (or transgender male person at birth)
* At least 18 years old
* HIV-seronegative
* Having had at least one anal sex episode with another man within the previous 6 months
* Having at least one of the following criteria:

  * Have a sexual partner (male or female) infected with HIV without evidence of virological suppression
  * Have had anal or vaginal sex episodes without condoms with more than one partner within the previous 6 months
  * Have had a sexually-transmitted infection (STI) within the previous 6 months (syndromic or biological approach, or mentioned by the participant)
  * Have received post-exposure prophylaxis for HIV within the previous 6 months
  * Wishing to reinforce its means of prevention through the use of PrEP
* Accepting to participate in the study and signing the informed consent form

Exclusion Criteria:

* Clinical manifestations suggesting a primary HIV infection
* Recent probable HIV exposure
* Creatinine clearance <60 mL/min calculated according to the Cockroft & Gault formula
* Positive or undetermined HBsAg
* Allergy or contraindication to any of the components of PrEP
* Participation in another biomedical and/or behavioral study on HIV or STIs (excluding CohMSM)
* Disability of the person making it difficult, if not impossible, to participate in the study or understanding of the information given to him
* Predictable non-compliance with the protocol (geographical distance, non-compliance with monitoring or other reasons)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of MSM under PrEP among eligible HIV-seronegative participants | 3 years
  To assess the acceptability of PrEP
Percentage of MSM using daily and/ord on-demand PrEP | 3 years
  To assess the acceptability of PrEP
Number of MSM followed after 3 years compared to the number of MSM included (retention in the program) | 3 years
  To assess the acceptability of PrEP
Percentage of adherence reported by MSM | 3 years
  To assess the adherence to PrEP
Counting of TDF/FTC tablets | 3 years
  To assess the adherence to PrEP
Plasma concentrations of TDF and FTC | 3 years
  To assess the adherence to PrEP
Percentage of HIV tests performed | 3 years
  To assess the adherence to quarterly HIV testing
Clinical and biological adverse events related to TDF and FTC | 3 years
  To assess the safety of daily and on-demand use of TDF/FTC
Frequency of condomless anal intercourse | 3 years
  To assess the evolution of the other prevention strategies on PrEP
Frequency of sexual intercourse associated with alcohol and/or drug use | 3 years
  To assess the evolution of the other prevention strategies on PrEP
Incidence rate of STIs | 3 years
  To assess the incidence of STIs on PrEP
Incidence rate of HIV infection | 3 years
  To assess the "real life" effectiveness of PrEP use and the emergence of treatment-related resistance
Percentage of TDF/FTC resistance among MSM newly infected by HIV | 3 years
  To assess the "real life" effectiveness of PrEP use and the emergence of treatment-related resistance
Total cost of the intervention over the study period and in the long term | 3 years
  To assess the cost and cost-effectiveness of PrEP
Incremental cost-effectiveness ratio of the intervention (versus no intervention) over the study period and in the long term | 3 years
  To assess the cost and cost-effectiveness of PrEP
Conditions of TDF/FTC price and of effectiveness for the intervention to be cost-effective in the study countries | 3 years
  To assess the cost and cost-effectiveness of PrEP

CONTACTS AND LOCATIONS:
Locations (4):
- Centre Oasis, Association African Solidarité, Ouagadougou, Burkina Faso
- Clinique de Confiance, Espace Confiance, Abidjan, Côte d’Ivoire
- Clinique des Halles, ARCAD-SIDA, Bamako, Mali
- Centre Lucia, Espoir Vie Togo, Lomé, Togo

REFERENCES:
- [Derived] Laurent C, Dembele Keita B, Yaya I, Le Guicher G, Sagaon-Teyssier L, Agboyibor MK, Coulibaly A, Traore I, Malan JB, De Baetselier I, Eubanks A, Riegel L, Rojas Castro D, Faye-Kette H, Kone A, Diande S, Dagnra CA, Serrano L, Diallo F, Mensah E, Dah TTE, Anoma C, Vuylsteke B, Spire B; CohMSM-PrEP Study Group. HIV pre-exposure prophylaxis for men who have sex with men in west Africa: a multicountry demonstration study. Lancet HIV. 2021 Jul;8(7):e420-e428. doi: 10.1016/S2352-3018(21)00005-9. Epub 2021 May 25. PMID 34048794